CLINICAL TRIAL: NCT03218865
Title: Evaluation of the Dialyzer Vitamin E Coated Effect Inflammatory State of Patients in ESRD and Its Clinical Benefits in Terms of Anemia
Brief Title: Influence of the Vitamine E Coated Dialyzer on Inflammation and Anemia
Acronym: EVIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hemotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EVIA 2012-A01502-41
Record Dates: First submitted 2017-07-04; First posted 2017-07-17 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: End Stage Renal Disease; Inflammation
MeSH Terms: conditions — Kidney Failure, Chronic; Inflammation

STUDY DESIGN:
Intervention Model Description: Prospective multicenter controlled and randomized protocol study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ViE High flux dialyzer (Experimental): vitamin E coated polysulfone membrane manufactured by Asahi Kasei Medical, with CE mark and intended for use in hemodialysis for the patient suffering from acute or chronic renal failure
  Interventions: Device: VIE high flux dialyzer
- Leoceed H high flux dialyzer (Active Comparator): polysulfone membrane manufactured by Asahi Kasei Medical, with CE mark and intended for use in hemodialysis for patient suffering from acute or chronic renal failure
  Interventions: Device: Leoceed H high flux dialyzer

INTERVENTIONS:
Device: VIE high flux dialyzer — Asssesment of the therapeutic effect of the vitamin E coating
  Arms: ViE High flux dialyzer
Device: Leoceed H high flux dialyzer — Use of the Leoceed H dialyzer during one year per patient enrolled in the control group
  Arms: Leoceed H high flux dialyzer

SUMMARY:
Evaluation of the effect of a vitamin E coated high flux polysulfone dialyzer on the inflammatory state of patients' end stage renal disease and its clinical benefits in terms of anemia Objectives : To assess the benefits of a vitamin E coated polysulfone membrane on the micro-inflammatory state of chronic dialysis patients Prospective multicenter controlled and randomized study Number of patients : 120 patients (60 patients per group)

DETAILED DESCRIPTION:
Coordinator : Pr JP.CRISTOL Montpellier hospital university Rational : The hemodialyzed patients are subject to inflammation due to their pathologies and to the technique. The VIE dialyzer polysulfon coated to vitamin E has been shown to have a favourable action on inflammation and anemia. The investigators want to highlight the influence of vitamine E graft using as controlled dialyzer a similar polysulfon from the same manufacturer without vitamin E.

Medical device : ViE High flux dialyzer -> vitamin E coated polysulfone membrane manufactured by Asahi Kasei Medical, with CE mark and intended for use in hemodialysis for the patient suffering from acute or chronic renal failure Controlled medical device : Leoceed H high flux dialyzer : polysulfone membrane manufactured by Asahi Kasei Medical, with CE mark and intended for use in hemodialysis for patient suffering from acute or chronic renal failure Objectives : To assess the benefits of a vitamin E coated polysulfone membrane on the micro-inflammatory state of chronic dialysis patients Primary end point : Evolution of the well-known inflammatory marker : High sensibility-CRP Secondary end point : Evolution of the following inflammatory markers : IL-6, TNFa, fibrinogen, antibodies anti- LDLox Evolution of Hemoglobin and ERI Evolution of Nutritional parameters : albumin and pre albumin Study design : Prospective multicenter controlled and randomized protocol study Duration : 12 months Number of patients : 120 patients : 60 patients per group 120 patients : 60 patients per group Adult ESRD patient, whatever the origin, treated by HD, thrice a week for about 4 hours and hemo dynamically well balanced Inclusion criteria : Dialyzed patient on synthetic high flux dialyzer for 3 months Patient with a vascular access allowing a blood flow rate ≥ 250 ml/min Patient with micro inflammation, i.e an average CRP between 5 and 20 mg/L on the two last check-up of CRP Patient informed of the study and having signed the inform consent. Exclusion criteria : Underage patient Subjects who are pregnant or planning to become pregnant during the study Patient with an infection influencing the Hb level

Patient with an Iron deficiency showed with :

Transferin saturation < 20 % and/or Ferritin < 100 µg/L, Hemo transfusion in the last two months Patient treated by HF, HDF, biofiltration Patient with infectious risks Subjects who participated in a clinical study involving dialyzers in the last two months

Criteria of exit :

Patient wish Medical decision Hemo transfusion Departure for another dialysis center Transplantation Death

ELIGIBILITY:
Inclusion Criteria:

* Adult ESRD patient, whatever the origin, treated by HD, thrice a week for about 4 hours and hemo dynamically well balanced
* Dialyzed patient on synthetic high flux dialyzer for 3 months
* Patient with a vascular access allowing a blood flow rate ≥ 250 ml/min
* Patient with micro inflammation, i.e an average CRP between 5 and 20 mg/L on the two last check-up of CRP
* Patient informed of the study and having signed the inform consent.

Exclusion Criteria:

* Underage patient
* Subjects who are pregnant or planning to become pregnant during the study
* Patient with an infection influencing the Hb level
* Patient with an Iron deficiency showed with :

Transferin saturation < 20 % and/or Ferritin < 100 µg/L,

* Patients having received an Hemo transfusion in the last two months
* Patient treated by HF, HDF, biofiltration
* Patient with infectious risks
* Subjects who participated in a clinical study involving dialyzers in the last two months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-10-16 (Actual); Primary Completion 2018-06-24 (Actual); Study Completion 2018-12-24 (Actual)

PRIMARY OUTCOMES:
Evolution of the well-known inflammatory marker : High sensibility-CRP | one year with a follow-up of three months
  Decrease of the CRP marker due the use of vitamin E coated dialyzer

SECONDARY OUTCOMES:
Inflammatory markers | one year with a follow-up of three months
  Evolution of the following inflammatory markers : IL-6, TNFalpha, fibrinogen, antibodies anti-LDLox
Anemia parameters | one year with a follow-up of three months
  Evolution of Hemoglobin and ERI
Nutritional Parameters | one year with a follow-up of three months
  Albumin and pre-albumin parameters

CONTACTS AND LOCATIONS:
Overall Officials: Jean Paul CRISTOL, Doctor, Study Director — AIDER association, clinique Jacques Mirouze 191 ave du Doyen Giraud 34295 Montpellier cedex 5
Locations (1):
- AIDER, Montpellier, Occitanie, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bargnoux AS, Cristol JP, Jaussent I, Chalabi L, Bories P, Dion JJ, Henri P, Delage M, Dupuy AM, Badiou S, Canaud B, Morena M. Vitamin E-coated polysulfone membrane improved red blood cell antioxidant status in hemodialysis patients. J Nephrol. 2013 May-Jun;26(3):556-63. doi: 10.5301/jn.5000195. Epub 2012 Sep 4. PMID 22956433